CLINICAL TRIAL: NCT06730204
Title: Nutrition Strategies and Malnutrition Assessment Management Systems for Preventing Malnutrition in Children With Solid Tumors: an Exploratory Intervention Study
Brief Title: Standardized Nutritional Management of Pediatric Patients With Solid Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: (2023)136
Record Dates: First submitted 2024-11-05; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Tumor, Solid; Children; Nutritional Intervention
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized nutrition management（+ short peptide ONS) Group (Experimental): The children in this group will be given standardized nutrition management after admission. They will follow the five-step treatment principle of malnutrition. Diet + nutrition education is the basic way, which is successively promoted to diet + oral nutrition supplement, enteral nutrition, partial enteral nutrition + supplementary parenteral nutrition, and total parenteral nutrition. When a nutritional treatment does not meet 60% of the target energy requirements for 3 to 5 days, the upper step of the treatment can be selected. For infants or newborns, when 75-80% of the target amount cannot be reached for 3-5 days, the upper step of the treatment can be selected.
  During the study period, an additional 3 months of short peptide oral nutritional supplements (ONS) is expected to be performed in children enrolled from December 1, 2024 to February 28, 2025 to explore the improvement of the nutritional status of the children.
  Interventions: Dietary Supplement: Standardized nutritional management; Dietary Supplement: Standardized nutritional management + short peptide ONS
- Control group (No Intervention): Clinical variables, biochemical markers, dietary data, and physical activity data will be collected at baseline and at each visit (admission to hospital, 1, 2, 3, 6, 12, 18, and 24 months after diagnosis).

INTERVENTIONS:
Dietary Supplement: Standardized nutritional management — The children will follow the five-step treatment principle of malnutrition. Diet + nutrition education is the basic way, which is successively promoted to diet + oral nutrition supplement, enteral nutrition, partial enteral nutrition + supplementary parenteral nutrition, and total parenteral nutrition. When a nutritional treatment does not meet 60% of the target energy requirements for 3 to 5 days, the upper step of the treatment can be selected. For infants or newborns, when 75-80% of the target amount cannot be reached for 3-5 days, the upper step of the treatment can be selected.
  Arms: Standardized nutrition management（+ short peptide ONS) Group
Dietary Supplement: Standardized nutritional management + short peptide ONS — During the study period, an additional 3 months of short peptide ONS enteral nutrition intervention is expected to be performed in children enrolled from Dec 1, 2024 to Feb 28, 2025 to explore the improvement of the nutritional status of the children. Short peptide type ONS 30ml/(kg.d) will be taken orally for children under 3 years old, and 20ml/(kg.d) for children over 3 years old. Due to conditional restrictions, standardized nutritional management + short peptide ONS intervention is only carried out in this subgroup.
  Inclusion criteria for short peptide ONS enteral nutrition intervention:
  1. Male and female, age 1-10 years old
  2. Pathological diagnosis is malignant solid tumor with untreated initial onset
  3. It is expected to receive enteral nutrition intervention for 3 months
  4. Clear consciousness, willing to cooperate, no serious dysfunction of major organ functions
  Arms: Standardized nutrition management（+ short peptide ONS) Group

SUMMARY:
The purpose of this study is to establish a standardized nutrition intervention procedure for children with solid tumors, and to explore the effectiveness and clinical applicability of standardized nutrition management and short peptide-based enteral nutrition intervention for improving the nutritional status of children with malignant solid tumors.

After admission, patients in the intervention group will receive standardized nutrition management provided by a nutrition support team composed of dietitians, nutritionists, clinicians, and nursing teams. Basic information, including diet, enteral and parenteral nutrition, nutritional status and clinical data, will be collected during the study.

ELIGIBILITY:
1. Male and female, age 0-18 years old
2. Pathological diagnosis is malignant solid tumor with untreated initial onset

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Weight for age Z score | 1, 2, 3, 6, 12, 18, and 24 months after enrollment
  Weight for age Z score = (Actual weight - reference population median) / reference population standard deviation
height/length for age Z score | 1, 2, 3, 6, 12, 18, and 24 months after enrollment
  Height/length for age Z score = (Actual height/length - reference population median) / reference population standard deviation
BMI for age Z score | 1, 2, 3, 6, 12, 18, and 24 months after enrollment
  BMI for age Z score = (Actual BMI - reference population median) / reference population standard deviation

SECONDARY OUTCOMES:
dietary intake | 1, 2, 3, 6, 12, 18, and 24 months after enrollment
  Unit: kcal/d A 24-hour dietary survey record will be conducted on the children to evaluate the quantity, type and energy of the food consumed.
serum albumin | 1, 2, 3, 6, 12, 18, and 24 months after enrollment
  Unit: g/L This indicator is measured by the biochemical assembly line Remisol in the hospital laboratory department.
serum prealbumin | 1, 2, 3, 6, 12, 18, and 24 months after enrollment
  Unit: mg/L This indicator is measured by the biochemical assembly line Remisol in the hospital laboratory department.
hemoglobin | 1, 2, 3, 6, 12, 18, and 24 months after enrollment
  Unit: g/L This indicator is measured by the hemocytometer XS800I in the hospital laboratory department.
electrolytes | 1, 2, 3, 6, 12, 18, and 24 months after enrollment
  Unit: mmol/L This indicator is measured by the biochemical assembly line Remisol in the hospital laboratory department.

OTHER OUTCOMES:
fecal intestinal flora | 3 months after enrollment
  For children with short peptide type enteral nutrition intervention, the above indicators will be collected at the time of enrollment and 3 months after enrollment.
Endotoxin | 3 months after enrollment
  For children with short peptide type enteral nutrition intervention, the above indicators will be collected at the time of enrollment and 3 months after enrollment.
Diamine oxidase | 3 months after enrollment
  For children with short peptide type enteral nutrition intervention, the above indicators will be collected at the time of enrollment and 3 months after enrollment.
D-lactic acid | 3 months after enrollment
  For children with short peptide type enteral nutrition intervention, the above indicators will be collected at the time of enrollment and 3 months after enrollment.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Olveira G, Tapia MJ, Ocon J, Cabrejas-Gomez C, Ballesteros-Pomar MD, Vidal-Casariego A, Arraiza-Irigoyen C, Olivares J, Conde-Garcia MC, Garcia-Manzanares A, Botella-Romero F, Quilez-Toboso RP, Matia P, Rubio MA, Chicharro L, Burgos R, Pujante P, Ferrer M, Zugasti A, Petrina E, Manjon L, Dieguez M, Carrera MJ, Vila-Bundo A, Urgeles JR, Aragon-Valera C, Sanchez-Vilar O, Breton I, Garcia-Peris P, Munoz-Garach A, Marquez E, Del Olmo D, Pereira JL, Tous MC. Hypoglycemia in noncritically ill patients receiving total parenteral nutrition: a multicenter study. (Study group on the problem of hyperglycemia in parenteral nutrition; Nutrition area of the Spanish Society of Endocrinology and Nutrition). Nutrition. 2015 Jan;31(1):58-63. doi: 10.1016/j.nut.2014.04.023. Epub 2014 May 10. PMID 25441588
- [Result] White JV, Guenter P, Jensen G, Malone A, Schofield M; Academy Malnutrition Work Group; A.S.P.E.N. Malnutrition Task Force; A.S.P.E.N. Board of Directors. Consensus statement: Academy of Nutrition and Dietetics and American Society for Parenteral and Enteral Nutrition: characteristics recommended for the identification and documentation of adult malnutrition (undernutrition). JPEN J Parenter Enteral Nutr. 2012 May;36(3):275-83. doi: 10.1177/0148607112440285. PMID 22535923
- [Result] Hulst JM, Zwart H, Hop WC, Joosten KF. Dutch national survey to test the STRONGkids nutritional risk screening tool in hospitalized children. Clin Nutr. 2010 Feb;29(1):106-11. doi: 10.1016/j.clnu.2009.07.006. Epub 2009 Aug 13. PMID 19682776
- [Result] Mohamed Elfadil O, Steien DB, Narasimhan R, Velapati SR, Epp L, Patel I, Patel J, Hurt RT, Mundi MS. Transition to peptide-based diet improved enteral nutrition tolerance and decreased healthcare utilization in pediatric home enteral nutrition. JPEN J Parenter Enteral Nutr. 2022 Mar;46(3):626-634. doi: 10.1002/jpen.2202. Epub 2021 Jul 19. PMID 34145597
- [Result] Leonard M, Caldari D, Mas E, Lambe C, Comte A, Ley D, Peretti N, Borderon C, Marinier E, Coste ME, Lamireau T, Rubio A, Turquet A, Dubern B, Dabadie A, Gautry J, Kyheng M, Guimber D, Gottrand F. Experience of Using a Semielemental Formula for Home Enteral Nutrition in Children: A Multicenter Cross-sectional Study. J Pediatr Gastroenterol Nutr. 2019 Apr;68(4):585-590. doi: 10.1097/MPG.0000000000002236. PMID 30896609
- [Result] Brinksma A, Sanderman R, Roodbol PF, Sulkers E, Burgerhof JG, de Bont ES, Tissing WJ. Malnutrition is associated with worse health-related quality of life in children with cancer. Support Care Cancer. 2015 Oct;23(10):3043-52. doi: 10.1007/s00520-015-2674-0. Epub 2015 Mar 10. PMID 25752883
- [Result] Becker P, Carney LN, Corkins MR, Monczka J, Smith E, Smith SE, Spear BA, White JV; Academy of Nutrition and Dietetics; American Society for Parenteral and Enteral Nutrition. Consensus statement of the Academy of Nutrition and Dietetics/American Society for Parenteral and Enteral Nutrition: indicators recommended for the identification and documentation of pediatric malnutrition (undernutrition). Nutr Clin Pract. 2015 Feb;30(1):147-61. doi: 10.1177/0884533614557642. Epub 2014 Nov 24. PMID 25422273
- [Result] Arends J, Bachmann P, Baracos V, Barthelemy N, Bertz H, Bozzetti F, Fearon K, Hutterer E, Isenring E, Kaasa S, Krznaric Z, Laird B, Larsson M, Laviano A, Muhlebach S, Muscaritoli M, Oldervoll L, Ravasco P, Solheim T, Strasser F, de van der Schueren M, Preiser JC. ESPEN guidelines on nutrition in cancer patients. Clin Nutr. 2017 Feb;36(1):11-48. doi: 10.1016/j.clnu.2016.07.015. Epub 2016 Aug 6. PMID 27637832
- [Result] Sasse P, Bergmann A, Afonso W, Ladas EJ, Ferman S. Malnutrition at diagnosis and throughout therapy in pediatric patients with solid tumors: A single-institution study in a developing country. Pediatr Blood Cancer. 2021 Nov;68(11):e29317. doi: 10.1002/pbc.29317. Epub 2021 Sep 7. PMID 34490992
- [Result] Runco DV, Stanek JR, Yeager ND, Belsky JA. Malnutrition identification and management variability: An administrative database study of children with solid tumors. JPEN J Parenter Enteral Nutr. 2022 Sep;46(7):1559-1567. doi: 10.1002/jpen.2329. Epub 2022 Feb 10. PMID 35040171
- [Result] Viana ECRM, Oliveira IDS, Rechinelli AB, Marques IL, Souza VF, Spexoto MCB, Pereira TSS, Guandalini VR. Malnutrition and nutrition impact symptoms (NIS) in surgical patients with cancer. PLoS One. 2020 Dec 15;15(12):e0241305. doi: 10.1371/journal.pone.0241305. eCollection 2020. PMID 33320857
- [Result] Bullock AF, Greenley SL, McKenzie GAG, Paton LW, Johnson MJ. Relationship between markers of malnutrition and clinical outcomes in older adults with cancer: systematic review, narrative synthesis and meta-analysis. Eur J Clin Nutr. 2020 Nov;74(11):1519-1535. doi: 10.1038/s41430-020-0629-0. Epub 2020 May 4. PMID 32366995
- [Result] Schoeman J. Nutritional assessment and intervention in a pediatric oncology unit. Indian J Cancer. 2015 Apr-Jun;52(2):186-90. doi: 10.4103/0019-509X.175832. PMID 26853397